CLINICAL TRIAL: NCT01942057
Title: Myopia Prevalence in Canadian School Children - a Pilot Study
Acronym: Falcon
Status: Completed | Type: Observational
Sponsor: University of Waterloo (Other)
Responsible Party: Sponsor
Other Study IDs: 19043
Record Dates: First submitted 2013-08-21; First posted 2013-09-13 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- School Grades 1+2: Children currently enrolled in grades 1 and 2
- School Grades 6+7: Children currently enrolled in grades 6 and 7
- School Grades 11+12: Children currently enrolled in grades 11 and 12

SUMMARY:
The goal of this study is to determine the prevalence of nearsightedness in Canadian school children living in the Waterloo Region.

ELIGIBILITY:
Inclusion Criteria:

* Has had a parent/legal guardian read the study consent form and who agrees to allow them to participate in the study by signing the consent form
* Has had the "letter of assent for children" explained to them, the child has agreed to participate and the letter has been signed by the study investigator and the child
* Has provided the completed Questionnaire (Appendix 4A for parents to complete on behalf of their children in school grades 1 and 2, 6 and 7; Appendix 4B for children to complete that are in school grades 11 and 12)
* Is currently in school grades 1 and 2, 6 and 7 or 11 and 12
* Is willing and able to follow instructions and maintain the appointment schedule

Exclusion Criteria:

* Has not given verbal assent to participate
* Has known sensitivity to the diagnostic pharmaceuticals to be used in the study
* Has undergone refractive error surgery or orthokeratology
* Has serious medical disorders or eye diseases/abnormalities such as amblyopia and cataract or a cognitive inability to conduct the tests

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: School children in Waterloo Region
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2013-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of children with spherical equivalent refraction of at least -0.50D in at least one eye | Day1

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, Principal Investigator — Center for Contact Lens Research
Locations (1):
- Centre for Contact Lens Research, Waterloo, Ontario, Canada

REFERENCES:
- See also: Centre for Contact Lens Research Website — http://cclr.uwaterloo.ca/